CLINICAL TRIAL: NCT07157319
Title: Zadek Osteotomy for Treatment of Haglund's Syndrome
Status: Recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mohamed Kamal Abdelhakeem, Orthopedics resident, Sohag University hospital, Sohag University
Other Study IDs: soh-Med--25-8-2MS
Record Dates: First submitted 2025-08-14; First posted 2025-09-05 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Haglund's Disease
Keywords: Zadek osteotomy for treatment of Haglund's syndrome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Haglund's syndrome is an abnormality of the bone and soft tissues in the foot. An enlargement of the bony section of the heel (where the Achilles tendon is inserted) triggers this condition.

* symptom includes insertional Achilles tendinopathy (IAT), The patient with HS often has a red, irritated, painful heel. And they often complain the enlargement of the posterior heel, which make it more difficult to footwear or sport
* Zadek described the Zadek Osteotomy option for the treatment of Haglund's syndrome This operation can change the calcaneus' anatomical length and elevate the distal insertion point of the Achilles tendon

  - It is a prospective case series study that will be done in Orthopedics and Traumatology department of Sohag university hospitals on patients suffering from Haglund's syndrome and treated by Zadek osteotomy
* This study aims to evaluate short term clinical, radiological and functional outcomes of Zadek osteotomy for treatment of Haglund's syndrome

DETAILED DESCRIPTION:
Introduction

* In 1928, Patrick Haglund described the Haglund syndrome firstly. Haglund's syndrome is an abnormality of the bone and soft tissues in the foot. An enlargement of the bony section of the heel (where the Achilles tendon is inserted) triggers this condition. The soft tissue near the back of the heel can become irritated when the large, bony lump rubs against rigid shoes.
* symptom includes insertional Achilles tendinopathy (IAT), The patient with HS often has a red, irritated, painful heel. And they often complain the enlargement of the posterior heel, which make it more difficult to footwear or sport.
* There are many conservative treatment options to treat it, which contains rest, activity modification, ice, or footwear modification.
* When these treatment for more than 6 months has failed, surgical options will be considered.
* Common surgical methods, including Haglund deformity debridement, endoscopic calcaneoplasty, and Zadek osteotomy (ZO).
* Zadek described the ZO option for the treatment of HS firstly. It was later modified by Keck and ZO is a dorsal closing wedge calcaneal osteotomy that allows the tuberosity of Haglund deformity to be brought forward. This operation can change the calcaneus' anatomical length and elevate the distal insertion point of the AT.

Aim of the work

• This study aims to evaluate short term clinical, radiological and functional outcomes of Zadek osteotomy for treatment of Haglund's syndrome.

Patients and Methods

* It is a prospective case series study that will be done in Orthopedics and Traumatology department of Sohag university hospitals on patients suffering from Haglund's syndrome and treated by Zadek osteotomy
* We are aiming in this study to include patients within period between 4/2025 to 10/2025

ELIGIBILITY:
Inclusion Criteria:

* patients over 18 years of age and less than 60 Yrs
* All patients had at least six months of conservative treatment

Exclusion Criteria:

1. patients below 18 years of age and more than 60 Yrs
2. patients of Haglund's syndrome with AT rupture or degeneration
3. uncontrolled diabetic patients with or without neuropathic joint destruction,
4. Infection such as osteomyelitis.
5. Charcot joint.
6. Peripheral vascular disease

Ages: 18 Years to 60 Years | Sex: All
Age Groups: Adult
Study Population: Patients attending and treating in Sohag University Hospital in Upper Egypt
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Primary outcomes for a Zadek osteotomy in Haglund's syndrome include: pain relief. | From enrollment and follow up to the end of 24 weeks
  - Pain Reduction: Marked improvement in pain, often measured by a Visual Analogue Scale (VAS) score, is a primary outcome, with significant reductions in pain intensity and frequency reported after the procedure.
functional improvement (measured by score VISA-A). | From enrollment and follow up to the end of 24 weeks
  Functional Improvement:
  VISA-A (Visual Analogue Scale for Achilles Tendinopathy) Score: A successful outcome is characterized by an improvement in the VISA-A score, reflecting better function for the Achilles tendon.
radiological changes to the calcaneus | From enrollment and follow up to the end of 24 weeks
  calcaneal length and tuberosity ratio (X/Y Ratio): The osteotomy modifies the calcaneus by shortening it and rotating the posterosuperior tuberosity, which reduces impingement on the Achilles tendon.
  calcaneal pitch angle(calcaneal inclination angle): Studies have shown a reduction in the calcaneal pitch angle after Zadek osteotomy which is a relevant radiological parameter for Haglund's deformity
improved ankle motion (dorsiflexion), | From enrollment and follow up to the end of 24 weeks
  Improvements in scores like the Tegner scale show a patient's ability to return to sports or other activities at a pre-injury level The Zadek osteotomy is known to improve the range of motion, specifically an increase in ankle dorsiflexion.
Patient Satisfaction: | From enrollment and follow up to the end of 24 weeks
  High rates of patient satisfaction are a key indicator of a successful procedure, with many patients reporting positive experiences post-surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of medicine, Sohag University, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided